CLINICAL TRIAL: NCT02118636
Title: Prospective Observational Study of Breast Cancer Patients Starting Therapy With an AI to Evaluate Mechanisms Underlying Development of Aromatase Inhibitor Associated Musculoskeletal Symptoms
Brief Title: Observational Study to Evaluate Mechanisms of Aromatase Inhibitor Associated Musculoskeletal Symptoms
Status: Completed | Type: Observational
Sponsor: Lynn Henry (Other)
Responsible Party: Sponsor-Investigator, Lynn Henry, Assistant Professor, University of Michigan Rogel Cancer Center
Organization: University of Michigan Rogel Cancer Center (Other)
Other Study IDs: UMCC 2009.057
Record Dates: First submitted 2014-01-15; First posted 2014-04-21 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer; Arthralgia
Keywords: Joint pain; Hormone receptor positive breast cancer; Estrogen; Androgen
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood is being collected at baseline for DNA extraction. Serum is being collected at baseline and after 3, 6, and 12 months.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aromatase inhibitor therapy: Subjects who are starting treatment with any of the three aromatase inhibitor (AI) medications

SUMMARY:
Early stage hormone receptor positive breast cancer is typically treated with adjuvant endocrine therapy in order to decrease risk of breast cancer recurrence and to improve overall survival from the disease. Typical agents used for treatment include tamoxifen and the aromatase inhibitors. In postmenopausal women, aromatase inhibitor therapy is increasingly common because it is associated with fewer long-term serious toxicities compared to tamoxifen. However, aromatase inhibitors cause arthralgias in 40-50% of patients, which can influence adherence to therapy and can lead to treatment discontinuation in a minority of cases. The mechanism underlying development of this toxicity remains unclear, and predictors of who will develop these symptoms remain undefined. This observational study is designed to collect patient-reported outcomes and serial serum samples in order to investigate potential etiologies of this bothersome toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer who are scheduled to receive endocrine therapy with an aromatase inhibitor
* All prior surgery, chemotherapy, and radiation therapy should be complete or should be completed by the time of AI treatment initiation (within 28 days of study enrollment)
* Age 21 and above and postmenopausal

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with hormone receptor positive breast cancer who are initiating therapy with an aromatase inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in estradiol and development of musculoskeletal symptoms between baseline and 3 months | 12 months
  To identify associations between estradiol serum concentrations at baseline and after 3 months of aromatase inhibitor therapy and the development of aromatase inhibitor-associated musculoskeletal symptoms by 12 months

SECONDARY OUTCOMES:
Change in sex hormones and development of musculoskeletal symptoms between baseline and 3 months | 12 months
  To identify associations between change in estrogens and androgens at baseline and 3 months of aromatase inhibitor therapy and development of aromatase inhibitor-associated musculoskeletal symptoms by 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States